CLINICAL TRIAL: NCT07339202
Title: Preoperative Hemodialysis Timing in Patients With End-Stage Kidney Disease: The POD-ESKD Pilot Trial
Acronym: POD-ESKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Vikram Fielding-Singh, Clinical Associate Professor, Department of Anesthesiology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69235; 5K23DK138312-02 (NIH)
Record Dates: First submitted 2026-01-12; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Perioperative Management; End Stage Kidney Disease (ESRD); Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Same-Day Hemodialysis (Experimental): Participants will receive same-day hemodialysis, defined as a hemodialysis treatment prior to the surgical procedure but on the same calendar day as the surgical procedure (typically in the morning prior to the procedure).
  Interventions: Procedure: Same-Day Hemodialysis
- No Same-Day Hemodialysis (Active Comparator): Participants will not receive same-day hemodialysis, defined as a hemodialysis treatment prior to the surgical procedure but on the same calendar day as the surgical procedure.
  Interventions: Procedure: No Same-Day Hemodialysis

INTERVENTIONS:
Procedure: Same-Day Hemodialysis — Hemodialysis treatment prior to the surgical procedure but on the same calendar day as the surgical procedure (typically in the morning prior to the procedure).
  Arms: Same-Day Hemodialysis
Procedure: No Same-Day Hemodialysis — No hemodialysis treatment prior to the surgical procedure but on the same calendar day as the surgical procedure.
  Arms: No Same-Day Hemodialysis

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of two different preoperative hemodialysis schedules for people with end-stage kidney disease (ESKD) who undergo surgical procedures. The main questions it aims to answer are:

Is it feasible to randomize participants with ESKD undergoing nonemergent surgical procedures to same-day hemodialysis versus no same-day hemodialysis?

Is it safe to randomize participants with ESKD undergoing nonemergent surgical procedures to same-day hemodialysis versus no same-day hemodialysis?

Researchers will compare the two hemodialysis schedules to see if the scheduling and safety profiles are the same.

Participants will:

Answer questions about their health up to 4 weeks before and 4 weeks after the surgical procedure.

Receive hemodialysis on the day of the surgical procedure or not, depending on the study treatment assignment.

DETAILED DESCRIPTION:
Participants will participate in the study for approximately 2 months, including assessment of 30-day postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing to comply with all study procedures for the duration of the study
2. Patient has a diagnosis of ESKD
3. Patient initiated hemodialysis at least 90 days prior to the planned surgical procedure
4. Patient is treated with a stable hemodialysis schedule, defined as an average of 2.5- 3.5 hemodialysis sessions per week in the preceding 4 weeks prior to surgery
5. Patient is scheduled to undergo nonemergent surgical procedures in the Stanford Health Care system. This includes (but is not limited to):

   * Fistula or graft creation, revision, or removal
   * Fistulogram
   * Peritoneal dialysis catheter placement or revision
   * Lower extremity angiogram (including femoral and iliac vessels)
   * Lower extremity bypass (including femoral and iliac vessels)
   * Lower extremity amputation
   * Lower extremity endarterectomy (including femoral and iliac vessels) Of note, this list of procedures is not exhaustive and other procedures may be considered that meet inclusion criteria and no exclusion criteria, in consultation with the treatment teams involved.

Exclusion Criteria:

1. Patient is pregnant
2. Patient is a prisoner
3. Patient is < 18 years old
4. The treating clinicians determine that the patient's clinical condition necessitate a specific approach to surgical scheduling or preoperative hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of hours from completion of the most recent preoperative hemodialysis session to entry into the operating room | up to 1 day
Number of participants who experience electrolyte abnormalities or volume overload requiring additional unplanned hemodialysis, rescheduling / cancellation of the surgical procedure, or an unanticipated escalation of postoperative level of care. | up to 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Fielding-Singh, MD, JD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fielding-Singh V, Vanneman MW, Grogan T, Neelankavil JP, Winkelmayer WC, Chang TI, Liu VX, Lin E. Association Between Preoperative Hemodialysis Timing and Postoperative Mortality in Patients With End-stage Kidney Disease. JAMA. 2022 Nov 8;328(18):1837-1848. doi: 10.1001/jama.2022.19626. PMID 36326747
- [Background] Fielding-Singh V, Vanneman MW, Morris AM, Winkelmayer WC, Sun LY, Roshanov PS, Montez-Rath ME, Chertow GM, Lin E. Preoperative Dialysis Dose and Postoperative Outcomes in Patients Receiving Maintenance Hemodialysis. Kidney360. 2025 Nov 1;6(11):1948-1959. doi: 10.34067/KID.0000000874. Epub 2025 Jun 12. PMID 40504620